CLINICAL TRIAL: NCT03419351
Title: Comparison of a Smartphone Based Self Refraction Tool With Conventional Refraction Error Estimation Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Martin Leitritz, Principal Investigator, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: smart-glass
Record Dates: First submitted 2017-12-06; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Refractive Errors; Self-Examination
MeSH Terms: conditions — Refractive Errors; Self-Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main group (Other): Main study group including all individuals that underwent the study procedures
  Interventions: Diagnostic Test: Smartphone; Diagnostic Test: Autorefractor; Diagnostic Test: Individual

INTERVENTIONS:
Diagnostic Test: Smartphone — Smartphone based measurement of refractive error and visual acuity testing using these measurements.
Diagnostic Test: Autorefractor — Autorefractor based measurement of refractive error and visual acuity testing using these measurements.
Diagnostic Test: Individual — Individual, human measurement of refractive error and visual acuity testing using these measurements.

SUMMARY:
Self evaluating tools based on smartphone devices are public available on the market for each person. The tools are used to estimate the existing refractive error for each eye of a patient. Hereafter, e.g. ordering glasses via internet could be the next step for this persons.

The daily routine within an eye hospital shows, that estimation of the refractive error is a difficult and time consuming procedure.

The study compares the results of the measured refractive error using a smartphone based tool with the results of conventional measurement methods.

ELIGIBILITY:
Inclusion Criteria:

* existing refractive error
* using glasses or contac lenses

Exclusion Criteria:

* opacities (visus limitating) of cornea, lens or vitreous
* known ocular pathologies except refractive error
* epilepsia
* irregular corneal topography

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Refractive Error | 6 month
  Comparison of refractive error measurements between methods

SECONDARY OUTCOMES:
Visual acuity | 6 month
  Visual acuity of persons using based on different methods.
Personal evaluation of measuring accuracy (Questionnaire) | 6 month
  Would persons be willing to order glasses by using only self-test-results?
Time consumption | 6 month
  Comparison of needed time to reach self-test refraction error results and conservative-test results.

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital, Tübingen, Baden-Wurttemberg, Germany